CLINICAL TRIAL: NCT07012278
Title: The Effect of St. John's Wort Oil on Wound Healing and Pain in Women Undergoing Cesarean Section: A Randomized Controlled Trial
Brief Title: St. John's Wort Oil for Wound Healing and Pain After Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, GÜLESER ADA, Research Assistant Dr., Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BARU-EBE-GA-02
Record Dates: First submitted 2025-05-30; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Wound Healing; Caesarean Section
Keywords: Caesarean section; wound healing; pain; St. John's wort oil
MeSH Terms: conditions — Pain | interventions — Hypericum extract LI 160

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): At the first follow-up, wound dressing will be performed using St. John's Wort oil, and participants will be instructed on how to apply the dressing themselves. They will be advised to apply the oil to the incision site once daily. With the participant's consent, photographs of the incision area will be taken.
  At the second follow-up, on postpartum day 15, the incision site will be evaluated by the researcher. With consent, photographs of the incision site will again be taken. Participants will be instructed to continue applying the oil daily.
  The third follow-up will take place on postpartum day 25, during which the REEDA Scale and the Numeric Rating Scale (NRS) will be administered to assess wound healing and pain.
  Interventions: Other: Caesarean section scar dressing with St. John's wort oil
- control (No Intervention): No intervention will be made to the control group. Only measurements will be made on parallel dates with the experimental group.

INTERVENTIONS:
Other: Caesarean section scar dressing with St. John's wort oil — Dressing the incision site with St. John's wort oil once a day every day
  Arms: Experimental group

SUMMARY:
Cesarean section refers to the surgical procedure in which the fetus is delivered via an incision, typically performed when vaginal delivery is not possible due to high-risk conditions. In recent years, the rate of cesarean deliveries has increased significantly. The quality of treatment and care is crucial in ensuring proper surgical wound healing following cesarean birth. Various new methods and products have been developed for wound healing and care in recent years, some of which are derived from herbal sources. The limitations of pharmacological methods used in the postpartum period, such as treatment failure, concerns about potential harm to the mother and infant, adverse side effects, negative impact on breastfeeding, emergence of resistant microorganisms, and ineffectiveness of current antibiotics, have led individuals to seek alternative natural remedies. Hypericum perforatum (commonly known as St. John's Wort) is frequently used in the postpartum period due to its antimicrobial and antioxidant properties. This study aims to examine the effects of Hypericum perforatum on wound healing and pain in women following cesarean delivery.

DETAILED DESCRIPTION:
Cesarean section is a surgical procedure in which the fetus is delivered through an incision when vaginal delivery is not possible due to certain high-risk conditions (1). In recent years, cesarean rates have increased rapidly, showing a 75% rise over the last 15 years (2). While the global cesarean rate was 7% in 1990, it has now reached 21% and is expected to continue increasing over the next decade. In Latin America and the Caribbean, 43% of all births are cesarean deliveries. In countries such as Egypt, Brazil, Cyprus, the Dominican Republic, and Turkey, cesarean births have surpassed vaginal deliveries (3).

Cesarean section is a life-saving intervention when maternal or fetal morbidity and mortality are at risk. However, due to the nature of the surgical procedure and anesthesia, cesarean delivery can lead to numerous physical and psychosocial problems during the postpartum period. One of the main factors negatively affecting infant care, mother-infant interaction, and the mother's ability to resume daily activities after cesarean delivery is the presence of a surgical wound. Delayed wound healing and wound-related complications are among the major issues encountered in the postpartum period (4). Approximately 5% of women who undergo cesarean delivery experience wound site complications such as hematoma, infection, and seroma (5).

A wound is defined as the disruption of the anatomical and functional integrity of intact skin and tissues due to trauma or surgical intervention (6,7). Wound healing is a critical process following cesarean delivery and is influenced by both local and systemic factors. Local factors include infection, oxygenation, necrotic tissue, foreign bodies, repeated trauma, and radiation exposure, while systemic factors encompass gender, chronic diseases, advanced age, immunodeficiency, nutritional deficiencies, smoking and alcohol use, obesity, medication use, and stress (8). Successful wound healing requires the orderly progression of distinct healing phases: hemostasis, inflammation, proliferation, and remodeling (5,6,8,9).

The quality of treatment and care plays a crucial role in the healing of surgical wounds after cesarean section (10). In recent years, new methods and products have been developed for wound care and healing, some of which are derived from herbal sources (9). Failures in pharmacological treatments applied in the postpartum period, concerns about the safety of these methods for the mother and infant, the presence of side effects, negative impacts on breastfeeding, the emergence of resistant microorganisms, and the inability of existing antibiotics to address these issues have all prompted individuals to seek natural alternatives (7,10,11,12).

These natural alternatives, collectively referred to as Traditional and Complementary Medicine (TCM), are defined by the World Health Organization (WHO) as "a set of knowledge, skills, and practices based on the theories, beliefs, and experiences indigenous to different cultures, used in the maintenance of health as well as in the prevention, diagnosis, improvement, or treatment of physical and mental illnesses" (13). TCM practices are widely used around the world. In China, they account for 40% of all medical treatments, and 80% of the population in Asia and Africa use TCM in primary healthcare services. In developed countries, 70% of the population in Canada, 75% in France, 42% in the USA, 30% in New Zealand, and 53% in Singapore report using TCM methods (7).

Herbal remedies are commonly used for wound care and healing. Globally, the use of medicinal plants accounts for approximately 60% of treatment approaches, with this rate ranging from 60% to 90% in developed countries (10). Herbs such as aloe vera, yarrow, hibiscus, chamomile, calendula, and St. John's wort are frequently utilized in wound healing due to their antioxidant, anticancer, antimicrobial, and anti-inflammatory properties. These plants also contribute to epithelialization, increased collagen synthesis, and enhanced fibroblast activity (7,10).

Hypericum perforatum (St. John's wort) is commonly used in the postpartum period because of its antimicrobial and antioxidant properties. A review of the literature shows that some studies have investigated the effects of St. John's wort oil on episiotomy wound care (14,15). However, no study has yet examined the effect of this oil on wound healing and pain following cesarean section. Therefore, this study aimed to evaluate the effects of Hypericum perforatum on wound healing and pain in women after cesarean delivery.

Study Design This study is planned as a true experimental, randomized controlled trial with a pretest-posttest design. The reporting of the study will adhere to the CONSORT (Consolidated Standards of Reporting Trials) guidelines. An application for registration will be submitted to ClinicalTrials.gov.

Sample Based on a power analysis conducted using G*Power 3.1.9.7, the required sample size was calculated to detect differences between groups with a Type I error of 0.05, a Type II error of 0.20, and an effect size of 0.70. Accordingly, 34 participants per group (a total of 68) were required. To account for potential dropouts, the sample size was increased by 15%, resulting in a planned total of 80 participants, with 40 assigned to each group.

Randomization Stratified block randomization will be used to assign participants to the intervention and control groups. Blocks will be repeated 20 times in each group (2x2x20), assigning a total of 80 participants in a balanced manner.

Data Collection Tools

The data will be collected using the following instruments:

Socio-Demographic Characteristics Form: Developed by the researchers, this form contains 18 questions to assess participants' socio-demographic and obstetric background.

REEDA Scale: Used to evaluate episiotomy and cesarean incision wounds. The scale was developed by Davidson (1970) and validated by Hill (1990). In Turkey, its validity and reliability were tested by Üstünsöz. The scale assesses five dimensions: Redness, Edema, Ecchymosis, Discharge, and Approximation. Each item is scored on a 4-point Likert scale (0-3), with total scores ranging from 0 to 15. Higher scores indicate poorer wound healing.

Numeric Rating Scale (NRS): This tool measures pain intensity on a numerical scale. It can be used in horizontal or vertical form and is typically rated from 0 (no pain) to 10 (worst possible pain).

Intervention: St. John's Wort Oil St. John's Wort oil (Hypericum perforatum) will be obtained from a certified manufacturer following Good Manufacturing Practices (GMP). The oil will be distributed to the participants in the intervention group.

Data Collection Period Data will be collected from women who agree to participate between June 30, 2025, and April 30, 2026. A total of 80 women will be included, consisting of 40 in the intervention group and 40 in the control group.

Inclusion Criteria Women who have undergone cesarean section and visit the Family Health Center within the first five days postpartum will be eligible for inclusion.

Follow-Up and Implementation

First follow-up (Day 5 postpartum): Participants in the intervention group will have their incision area dressed with St. John's Wort oil. Instructions on how to self-administer the dressing once daily will be provided. With consent, photographs of the incision area will be taken.

Second follow-up (Day 15 postpartum): The wound site will be evaluated by the researcher. Photographs will again be taken with consent, and participants will be advised to continue using the oil.

Third follow-up (Day 25 postpartum): Both the REEDA Scale and the NRS will be administered to assess wound healing and pain.

Control Group Protocol Participants in the control group will not receive any intervention. Their incision sites will be photographed during the second and third follow-ups (with consent), and the REEDA and NRS scales will be applied during the first and final assessments.

Target Sample Size A total of 80 participants, 40 in the intervention group and 40 in the control group, will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Having had a cesarean section,
* Her first cesarean section,
* Being fluent in Turkish.

Exclusion Criteria:

* Not wanting to participate in the research,
* The existence of a communication barrier.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
pre-test post-test | 6 months
  In the first follow-up, a dressing will be made with St. John's wort oil and the woman will be told how to make a dressing with this oil. It will be explained to the woman to make a dressing with St. John's wort oil at the incision site once a day every day. The incision site will be photographed for women who give permission.
pre-test post-test | 6 months
  On the 15th day, which is the second follow-up, the wound site will be evaluated by the researcher. The incision site of the women who give permission will be photographed. She will be told to continue the application of St. John's wort oil.
pre-test post-test | 6 months
  The third follow-up will be performed on the 25th postpartum day. REEDA Scale and NRS Scale will be applied. REEDA Scale: REEDA scale is used in the evaluation of episiotomy and cesarean incision wounds. The REEDA scale was developed by Davidson in 1970 and used in his master's thesis on the monitoring of wound healing in the perineum. The validity and reliability study of the scale was conducted by Hill in 1990. In Turkey, the validity and reliability study of the REEDA Scale was conducted by Üstünsöz and used in her master's thesis titled "The Effect of Hot and Cold Applications in Episiotomy Healing". The scale has five sub-dimensions: redness, edema, ecchymosis, discharge and approximation of wound edges. Each sub-dimension of the scale is graded using a 4 (four) point Likert-type rating. The evaluation is made between 0-3. The sum of the scale score varies between 0-15. The higher the scale score, the worse the wound healing.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Nur Yıldırım Bayraktar, PhD, Study Chair — sakarya üniversity; Kevser İLÇİOĞLU Associate Professor, PhD, Study Director — sakarya üniversity
Locations (1):
- Sakarya Üniversity, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No